CLINICAL TRIAL: NCT03929497
Title: Interventional, Open-label, Flexible-dose, Long-term Safety Extension Study of Lu AF11167 in Patients With Schizophrenia
Brief Title: Flexible-dose Long-term Extension Study of Lu AF11167 in Patients With Schizophrenia With Prominent Negative Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy based on the interim analysis in the 17972A study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17972B
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF11167 (Experimental)
  Interventions: Drug: Lu AF11167

INTERVENTIONS:
Drug: Lu AF11167 — Lu AF11167 - 2 or 4 mg/day; tablets, orally

SUMMARY:
A study to evaluate the long-term safety and tolerability of flexible doses of Lu AF11167 in patients with schizophrenia during the 24-week treatment period

ELIGIBILITY:
Inclusion Criteria:

* The patient completed Study 17972A.
* The patient and the patient's caregiver or identified responsible person is able to read and understand the Informed Consent Form.
* The patient has signed the Informed Consent Form specific for Study 17972B.
* The patient can potentially benefit from 24 weeks of treatment with Lu AF11167 according to the investigator's clinical judgment.

Exclusion Criteria:

* The patient has any current primary psychiatric disorder other than schizophrenia diagnosed during study 17972A
* The patient, in the opinion of the investigator, is at significant risk of suicide

Other in- and exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events | From baseline week 24
  Safety and Tolerability based on the safety assessments (clinical safety laboratory tests, vital signs, BMI, waist, weight, ECG parameters)

SECONDARY OUTCOMES:
Change in Brief Negative Symptom Scale (BNSS) total score | from baseline to Week 24
  The BNSS is a brief clinician rating scale, intended to measure negative symptoms. It consists of 13 items organized into 6 subscales: anhedonia, distress, asociality, avolition, blunted affect, and alogia. The items score the impairment. Items 1 to 4 are rated from 0 (Normal) to 6 (Extremely severe) and items 5 to 13 are rated from 0 (No impairment) to 6 (Severe deficit). The BNSS total score is calculated by summing the 13 individual items; subscale scores are calculated by summing the individual items within each subscale. Users of the BNSS should have training in psychiatric interview techniques and have clinical experience working with patients with schizophrenia and related psychotic disorders. The BNSS total scores ranges from 0 to 78.
Change in Positive and Negative Syndrome Scale (PANSS) Marder Negative Symptoms Factor Score | from baseline to Week 24
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items: 7 items make up the positive scale (for example: delusions, conceptual disorganization and hallucinatory behaviour), 7 items make up the negative scale (for example: blunted affect, emotional withdrawal and poor rapport) and 16 items make up the general psychopathology scale (for example: somatic concern, anxiety and guilt feelings). Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). The PANSS total score is the sum of all items, and ranges from 30 to 210. Subscale scores are the sum of items within each subscale.
Change in PANSS Negative subscale score | from baseline to Week 24
  The PANSS is a clinician rated scale designed to measure severity of psychopathology in adult patients with schizophrenia, schizoaffective disorders and other psychotic disorders. It emphasizes positive and negative symptoms. The PANSS includes 3 sub-scales and 30 items: 7 items make up the positive scale (for example: delusions, conceptual disorganization and hallucinatory behaviour), 7 items make up the negative scale (for example: blunted affect, emotional withdrawal and poor rapport) and 16 items make up the general psychopathology scale (for example: somatic concern, anxiety and guilt feelings). Each item is rated from 1 (symptom not present) to 7 (symptom extremely severe). The PANSS total score is the sum of all items, and ranges from 30 to 210. Subscale scores are the sum of items within each subscale.
Change in CGI-SCH-S negative symptoms score | from baseline to Week 24
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive, and depressive) and the overall severity of the disorder. The CGI-SCH-severity of illness symptoms and overall severity are rated on a 7-point scale ranging from 1 (normal - not ill) to 7 (Among the most severely ill). For the first four ratings (positive, negative, depressive, and cognitive symptoms), the assessment should focus on the severity of symptoms only. Additionally, for 'overall severity' rating, both severity of symptoms and interference with functioning should be considered.
CGI-SCH-DC negative symptoms score | at Week 24
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive, and depressive) and the overall severity of the disorder. The CGI-SCH-degree of change symptoms and overall severity are rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Each single rating (conditions of severity and degree of change) and overall ratings of severity and improvement are scored independently and no total score is derived.
CGI-SCH-DC negative symptoms response | at Week 24
  The CGI-SCH is a clinician-rated scale to assess global illness severity and degree of change in patients with schizophrenia. For both the global illness severity and degree of change, the CGI-SCH consists of four different groups of symptoms (positive, negative, cognitive, and depressive) and the overall severity of the disorder. The CGI-SCH-degree of change symptoms and overall severity are rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Each single rating (conditions of severity and degree of change) and overall ratings of severity and improvement are scored independently and no total score is derived.CGI-SCH-DC negative symptoms response is defined as a CGI-SCH-DC negative symptoms score of 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (30):
- Bulgaria (10):
  - Mental Health Center Prof. Dr. Ivan Temkov EOOD (BG0001), Burgas
  - MHAT Dr. Hristo Stambolski (BG0007), Kazanlak
  - First Department for men with acute mental diseases-NPH Sv. Ivan Rilski (BG0010), Novi Iskar
  - UMHAT Dr.Georgi Stranski EAD (BG0006), Pleven
  - State Psychiatric Hospital - Sevlievo (BG0009), Sevlievo
  - Medical Center INTERMEDICA (BG0003), Sofia
  - DCC Mladost-M (BG0004), Varna
  - Med Centre Medical plus (BG0008), Varna
  - DCC Mladost-M Varna OOD (BG0005), Varna
  - Mental Health Center-Vratsa EOOD (BG0002), Vratsa
- Estonia (2):
  - Marienthali Kliinik (EE0001), Tallinn
  - OU Jaanson & Laane (EE0002), Tartu
- Office of Dr.Kirsten Hahn MD (DE0002), Berlin, Germany
- Hungary (4):
  - Semmelweis Egyetem Neurologiai Klinika-Semmelweis University (HU0005), Budapest
  - Bugat Pal Hospital (HU0008), Gyöngyös
  - Dr Mathe es Tarsa Bt (HU0001), Kalocsa
  - Javorszky Odon Hospital (HU0004), Vác
- Latvia (3):
  - Hospital Gintermuiza (LV0001), Jelgava
  - Riga Centre Of Psychiatry And Addiction Disorders (LV0002), Riga
  - Sigulda Hospital Outpatient Clinic (LV0006), Sigulda
- Syntonia Sp. z o.o. (PL0002), Pruszcz Gdański, Poland
- Ukraine (9):
  - Si Inpn Namsu (Ua0003), Kharkiv
  - Si Inpn Namsu (Ua0008), Kharkiv
  - Kherson Regional Psychiatric Hospital (UA0009), Kherson
  - Kiev Regional Specialized Psycho-Narcological Medical Care (UA0005), Kiev
  - Regional Clinical Psychiatry Hospital of Kirovograd Regional Council, Donetsk National Medical University (UA0004), Kropyvnytskyi
  - "Kyiv Railway Clinical Hospital ¿1 of Branch ""Health Center"" of the Public joint stock company ""Ukrainian Railway"", psychoneurological department" (UA0007), Kyiv
  - Odessa Regional Medical Centre of Mental Health (UA0006), Odesa
  - Ukrainian Medical Stomatological Academy (UA0001), Poltava
  - Vinnitsa National Medical University (UA0002), Vinnytsia

REFERENCES:
- [Derived] Meyer-Lindenberg A, Nielsen J, Such P, Lemming OM, Zambori J, Buller R, der Goltz CV. A double-blind, randomized, placebo-controlled proof of concept study of the efficacy and safety of Lu AF11167 for persistent negative symptoms in people with schizophrenia. Eur Neuropsychopharmacol. 2022 Aug;61:4-14. doi: 10.1016/j.euroneuro.2022.05.009. Epub 2022 Jun 12. PMID 35704951